CLINICAL TRIAL: NCT00285636
Title: Long Term Follow-Up of Burn Injuries
Status: Completed | Type: Observational
Sponsor: National Institutes of Health (NIH) (NIH)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, David R. Patterson, Professor, National Institute of General Medical Sciences (NIGMS)
Organization: National Institute of General Medical Sciences (NIGMS) (NIH)
Other Study IDs: 95-0217-C; 97-4938-C08
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2009-09

CONDITIONS: Burn
Keywords: Long Term Follow-Up
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to investigate the psychological effects of burn injuries as experienced by patients.

DETAILED DESCRIPTION:
We are interested in determining how people adjust to burn injuries as a way of facilitating optimal recovery. This is done by conducting several questionnaires at the time of the discharge in the hospital, and later follow up with the patients up to two years.

ELIGIBILITY:
Inclusion Criteria:

* patients with more than a 30% total surface area burn
* English speaking

Exclusion Criteria:

* Patients with less than a 30% total surface area burn
* Non English speaking

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: burn patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 1992-06; Primary Completion 2007-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Patterson, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington; Harborview Medical Center, Seattle, Washington, United States